CLINICAL TRIAL: NCT02526628
Title: The Haemostatic Balance and Neurocognitive Phenotype in Klinefelter Syndrome - The Effect of Testosterone Treatment
Brief Title: Thrombosis and Neurocognition in Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); University of Southern Denmark (Other); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_KS_TESTOSTERONE
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2018-01

CONDITIONS: Klinefelter Syndrome; Thrombosis
Keywords: Testosterone; Neurocognition
MeSH Terms: conditions — Klinefelter Syndrome; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Bloodsamples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Testosterone naïve KS: Men with Klinefelter syndrome without testosterone treatment. After initial examination standard treatment with testosterone will be effectuated according to current guidelines.
- Testosterone treated KS: Men with Klinefelter syndrome receiving testosterone treatment
- Controls 1: Matched healthy male controls for testosterone naive KS
- Controls 2: Matched healthy male controls for testosterone treated KS

SUMMARY:
The haemostatic balance and neurocognitive capability of men with Klinefelter syndrome is compared to healthy controls by using specific biochemical assays for coagulation and fibrinolysis and a selection of neuropsychological tests and brain fMRI. Furthermore, the effect of gonadal status and any effects of long- or short-term testosterone treatment on the above mentioned parameters are investigated.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS) affects approximately 1 in every 600 males, but remains severely underdiagnosed. Men with KS are more prone to a wide range of diseases including thrombotic disorders. Also, neurocognitive function is impaired in KS. The background for the increased thrombosis proneness is not understood, and also it is not understood how testosterone treatment affects the thrombosis risk in KS. The effects of testosterone treatment on neurocognition in KS is also not completely understood. However, it is speculated that testosterone treatment at an early point could help improve the overall neurocognitive performance.

In this study 30 males with KS receiving testosterone treatment, 30 males with KS not receiving testosterone treatment and 60 matched healthy male controls are included. After initial examination including blood testing and neurocognitive testing, the subjects are followed for 18 months and examined a second time. After initial examination the group of previously untreated KS males will be put on standard testosterone treatment according to current guidelines.

Groups will be compared by measuring and array of markers for coagulation and fibrinolysis, including thrombin generation and fibrin structure analysis, to assess the haemostatic balance. Also, a wide array of neurocognitive tests and brain fMRI is applied to compare the neurocognitive function between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter syndrome with 47 XXY karyotype
* Healthy male

Exclusion Criteria:

* Known thrombophilia
* Previous thrombotic event
* Chronic or acute illness affecting the haemostatic balance (e.g. diabetes, cancer).
* Previous or current disease affecting the brain
* Weight above 120 kg
* Current abuse of stimulants affecting the brain
* Unability to complete MR-scan (e.g. claustrophobia, internal metal objects)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with Klinefelter syndrome identified through clinics for fertility, endocrinology and genetics. Healthy controls from the general population living in Central Denmark Region.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-09; Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Differences in thrombin generation | Time 0 and after 18 months followup
  Thrombin generation using the CAT assay is assessed as ETP (nM thrombin), peak height (nM thrombin) and lag time (minutes). All variables are assessed at inclusion and after a 18 month follow-up. Groups are compared statistically at each time point and any changes during follow-up is also analysed.
Differences in fibrin clot properties | Time 0 and after 18 months followup
  Fibrin clot properties is assessed by fibrin structure analysis in plasma samples. All variables are assessed at inclusion and after a 18 month follow-up. Groups are compared statistically at each time point and any changes during follow-up is also analysed.
Difference in neurocognition | Time 0 and after 18 months followup
  neurocognition is assessed using a wide array of psychological tests (e.g. Wais-III, Stroop test, Wisconsin Card Sorting Test and others) All variables are assessed at inclusion and after a 18 month follow-up. Groups are compared statistically at each time point and any changes during follow-up is also analysed.

SECONDARY OUTCOMES:
Differences in blood coagulation and fibrinolysis parameters between groups | Time 0 and after 18 months followup
  Coagulation and fibrinolysis can not be adequately assessed by analysis of a single parameter. To evaluate the overall status of these systems an array of analyses are needed, and further more need to be interpreted by experts within the field. Thus, severeal markers of coagulation and fibrinolysis including INR, APTT, single coagulation factors, PAI-1 and others are to be assessed at inclusion and after a 18 month follow-up. Groups are compared statistically at each time point and any changes during follow-up is also analysed. Besides applying statistics, the compiled results will also be interpreted by experts within the field to provide an overall characterization of the haemostatic balance in the individual groups and by comparison to each other.
Differences in fMRI between groups | Once at followup
  fMRI will be performed to evaluate the response in the brain to various stimuli and tests, with the overall purpose of examining speech, memory and other cognition related features.

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, MD, Prof., Study Chair — Department of Endocrinology and Internal Medine and Department of Molecular Medicine; Simon Chang, MD, Principal Investigator — Unit for Thrombosis Research; Anne Skakkebæk, MD, PhD, Principal Investigator — Department of Clinical Genetics
Locations (1):
- Department for Endocrinology and Internal Medicine, Aarhus, Denmark

REFERENCES:
- [Derived] Viuff M, Skakkebaek A, Johannsen EB, Chang S, Pedersen SB, Lauritsen KM, Pedersen MGB, Trolle C, Just J, Gravholt CH. X chromosome dosage and the genetic impact across human tissues. Genome Med. 2023 Mar 28;15(1):21. doi: 10.1186/s13073-023-01169-4. PMID 36978128